CLINICAL TRIAL: NCT04711239
Title: Non-invasive Preimplantation Genetic Testing for Aneuploidies (niPGT-A) - Evaluation of the Analysis of Cell-free DNA in Spent Culture Medium
Brief Title: Non-invasive Preimplantation Genetic Testing for Aneuploidies Using Cell-free DNA in Spent Culture Media
Acronym: niPGT-A
Status: Withdrawn | Type: Observational
Why Stopped: Unavailability of Primary investigator
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-ABU-011-SJ
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Secondary Infertility
Keywords: PGT-A; cell-free DNA; spent culture media; NGS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples to be collected:
  * Saliva sample from female patient for maternal DNA contamination assessment
  * Spent culture media (SCM) collected on the day of biopsy
  * Trophectoderm (TE) biopsy for clinical PGT-A
  All samples collected for the study will be labelled with anonymised sample identifiers and cryopreserved until time of analysis. SCM samples will be stored at -80°C and TE biopsies at -20°C. Saliva samples will be stored at room temperature prior to DNA extraction. Extracted/amplified DNA will be stored at 4°C until completion of analysis, then at -20°C.
  Once the study is finalised, all stored samples will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two types of samples (TE and SCM) will be collected for all blastocysts included in the study
  Interventions: Diagnostic Test: PGT-A / niPGT-A

INTERVENTIONS:
Diagnostic Test: PGT-A / niPGT-A — PGT-A and niPGT-A will be performed using next generation sequencing (NGS) analysis for chromosome copy number variation (CNV). Embryo transfers will rely solely on the results of PGT-A for trophectoderm biopsies.

SUMMARY:
Analysis of embryonic cell-free DNA (cfDNA) present in the spent culture media (SCM) is a non-invasive alternative for preimplantation genetic testing for aneuploidies (PGT-A) that avoids the technical challenges and limitations of biopsy. Initial studies investigating this non-invasive PGT-A (niPGT-A) method reported variable concordance between cfDNA in SCM and the trophectoderm sample (~ 30%-86%) and indicated a contribution from both the inner cell mass and trophectoderm to the cfDNA in SCM.

This study aims to evaluate the use of the embryo culture medium as a source of genetic material for PGT-A and validate a niPGT-A protocol using cfDNA in SCM.

DETAILED DESCRIPTION:
Multiple studies have demonstrated the ability to detect and amplify cfDNA from SCM, at different stages of embryonic development, with varying rates of amplification success. Differences in analytes, timing of SCM collection and the duration of embryo culture within the collected medium, performance of assisted hatching (AH), whole genome amplification methods, comprehensive chromosome screening methods and next generation sequencing (NGS) platforms, bioinformatic analyses and strategies for identifying maternal contamination all contribute to the ultimate performance of niPGT-A.

This study aims to validate a noninvasive PGT-A (niPGT-A) method utilizing cfDNA released from the human blastocyst into the SCM.

Patients undergoing a fertility treatment with PGT-A due to secondary infertility will be recruited. On day 6 post fertilization, SCM will be collected prior to blastocyst biopsy. The SCM is normally discarded at this stage. Trophectoderm biopsy and sample collection will follow the IVF laboratory's standard practices for clinical PGT-A.

Three aneuploidy screening kits, relying on different whole genome amplification methods followed by NGS on the Ion GeneStudio™ S5 Prime System (ThermoFisher Scientific), will be compared. The concordance between cfDNA and trophectoderm biopsies will be evaluated for approximately 150 blastocysts with the best performing niPGT-A protocol.

Selection of the embryo(s) for transfer will be based solely on the PGT-A result from the biopsied cells. The patient's IVF+PGT-A treatment plan and timeline will not be altered.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fertility treatment with PGT-A (Recombinant FSH antagonist protocol with dual trigger)
* Secondary infertility
* BMI 18- 35 kg/m2
* Sperm: fresh ejaculated sperm (abstinence: 2-3 days)
* At least one blastocyst biopsied on day 6

Exclusion Criteria:

* High progesterone on day of trigger (>1.5ng/ml)
* Vitrified oocytes
* Frozen sperm
* Indications for PGT-SR and PGT-M

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Day 6 blastocysts generated from couples undergoing fertility treatment with PGT-A and meeting the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
General concordance between results for cfDNA in SCM and trophectoderm biopsies | 4 months
  General ploidy concordance rate: number of matched (euploid-euploid or aneuploid-aneuploid) result/total number cfDNA samples with a result
Discordance per chromosome between results for cfDNA in SCM and trophectoderm biopsies | 4 months
  Discordance per chromosome: number of misidentified chromosomal errors/24*total number of embryos with cfDNA result
Concordance per chromosome between results for cfDNA in SCM and trophectoderm | 4 months
  Chromosome error concordance: number of correctly identified chromosomal errors/total number of chromosomal errors detected
Sensitivity of niPGT-A using cfDNA in SCM | 4 months
  False negative rate: 1- (true euploid result/total number of samples with a result)
Specificity of niPGT-A using cfDNA in SCM | 4 months
  False positive rate: 1- (true aneuploid result/total number of samples with a result)

SECONDARY OUTCOMES:
Pregnancy outcome for patients having an embryo transfer - Implantation rate | 12 months
  Implantation rate = number of gestational sacs observed at echographic screening at 6 weeks of pregnancy / number of embryos transferred
Pregnancy outcome for patients having an embryo transfer - Biochemical pregnancy rate | 12 months
  Biochemical pregnancy rate = positive βhCG test of > 15IU but no foetal heartbeat / gestational sac on ultrasound examination
Pregnancy outcome for patients having an embryo transfer - Clinical pregnancy rate | 12 months
  Clinical pregnancy rate (%) defined by positive βhCG test and ultrasound confirmation of gestational sac or heartbeat
Pregnancy outcome for patients having an embryo transfer - Miscarriage rate | 12 months
  Miscarriage rate (%) defined by ultrasonographic visualization of one or more gestational sacs, including ectopic pregnancies, with spontaneous pregnancy loss prior to 20 weeks
Pregnancy outcome for patients having an embryo transfer - Clinical pregnancy rate | 12 months
  Ongoing pregnancy rate (beyond 20 weeks)
Pregnancy outcome for patients having an embryo transfer - Implantation failure rate | 12 months
  Implantation Failure (%)

CONTACTS AND LOCATIONS:
Overall Officials: Souraya Jaroudi, Principal Investigator — ART Fertility Clinics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shamonki MI, Jin H, Haimowitz Z, Liu L. Proof of concept: preimplantation genetic screening without embryo biopsy through analysis of cell-free DNA in spent embryo culture media. Fertil Steril. 2016 Nov;106(6):1312-1318. doi: 10.1016/j.fertnstert.2016.07.1112. Epub 2016 Aug 24. PMID 27565258
- [Background] Xu J, Fang R, Chen L, Chen D, Xiao JP, Yang W, Wang H, Song X, Ma T, Bo S, Shi C, Ren J, Huang L, Cai LY, Yao B, Xie XS, Lu S. Noninvasive chromosome screening of human embryos by genome sequencing of embryo culture medium for in vitro fertilization. Proc Natl Acad Sci U S A. 2016 Oct 18;113(42):11907-11912. doi: 10.1073/pnas.1613294113. Epub 2016 Sep 29. PMID 27688762
- [Background] Feichtinger M, Vaccari E, Carli L, Wallner E, Madel U, Figl K, Palini S, Feichtinger W. Non-invasive preimplantation genetic screening using array comparative genomic hybridization on spent culture media: a proof-of-concept pilot study. Reprod Biomed Online. 2017 Jun;34(6):583-589. doi: 10.1016/j.rbmo.2017.03.015. Epub 2017 Mar 28. PMID 28416168
- [Background] Rubio C, Navarro-Sanchez L, Garcia-Pascual CM, Ocali O, Cimadomo D, Venier W, Barroso G, Kopcow L, Bahceci M, Kulmann MIR, Lopez L, De la Fuente E, Navarro R, Valbuena D, Sakkas D, Rienzi L, Simon C. Multicenter prospective study of concordance between embryonic cell-free DNA and trophectoderm biopsies from 1301 human blastocysts. Am J Obstet Gynecol. 2020 Nov;223(5):751.e1-751.e13. doi: 10.1016/j.ajog.2020.04.035. Epub 2020 May 26. PMID 32470458
- [Background] Fang R, Yang W, Zhao X, Xiong F, Guo C, Xiao J, Chen L, Song X, Wang H, Chen J, Xiao X, Yao B, Cai LY. Chromosome screening using culture medium of embryos fertilised in vitro: a pilot clinical study. J Transl Med. 2019 Mar 8;17(1):73. doi: 10.1186/s12967-019-1827-1. PMID 30849973
- [Background] Huang L, Bogale B, Tang Y, Lu S, Xie XS, Racowsky C. Noninvasive preimplantation genetic testing for aneuploidy in spent medium may be more reliable than trophectoderm biopsy. Proc Natl Acad Sci U S A. 2019 Jul 9;116(28):14105-14112. doi: 10.1073/pnas.1907472116. Epub 2019 Jun 24. PMID 31235575
- [Background] Capalbo A, Romanelli V, Patassini C, Poli M, Girardi L, Giancani A, Stoppa M, Cimadomo D, Ubaldi FM, Rienzi L. Diagnostic efficacy of blastocoel fluid and spent media as sources of DNA for preimplantation genetic testing in standard clinical conditions. Fertil Steril. 2018 Oct;110(5):870-879.e5. doi: 10.1016/j.fertnstert.2018.05.031. PMID 30316433
- [Background] Ho JR, Arrach N, Rhodes-Long K, Ahmady A, Ingles S, Chung K, Bendikson KA, Paulson RJ, McGinnis LK. Pushing the limits of detection: investigation of cell-free DNA for aneuploidy screening in embryos. Fertil Steril. 2018 Aug;110(3):467-475.e2. doi: 10.1016/j.fertnstert.2018.03.036. Epub 2018 Jun 28. PMID 29960707
- [Background] Kuznyetsov V, Madjunkova S, Antes R, Abramov R, Motamedi G, Ibarrientos Z, Librach C. Evaluation of a novel non-invasive preimplantation genetic screening approach. PLoS One. 2018 May 10;13(5):e0197262. doi: 10.1371/journal.pone.0197262. eCollection 2018. PMID 29746572
- [Background] Vera-Rodriguez M, Diez-Juan A, Jimenez-Almazan J, Martinez S, Navarro R, Peinado V, Mercader A, Meseguer M, Blesa D, Moreno I, Valbuena D, Rubio C, Simon C. Origin and composition of cell-free DNA in spent medium from human embryo culture during preimplantation development. Hum Reprod. 2018 Apr 1;33(4):745-756. doi: 10.1093/humrep/dey028. PMID 29471395